CLINICAL TRIAL: NCT06378268
Title: Effectiveness of Progestin-Primed Ovarian Stimulation Versus GnRH Antagonist Protocol for Ovarian Stimulation in IVF: a Randomized Clinical Trial
Brief Title: PPOS vs GnRH Antagonist in Ovarian Stimulation (ProGanOS Study)
Acronym: ProGanOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/24/DD-BVMD
Record Dates: First submitted 2024-04-07; First posted 2024-04-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Progestins Primed Ovarian Stimulation
Keywords: Progestins Primed Ovarian Stimulation; GnRH antagonist; ongoing pregnancy
MeSH Terms: interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Progestins Primed Ovarian stimulation group (Active Comparator): PPOS group: Recombinant FSH 150-300 IU/day will start from day 2 to day 4 of menstruation. The initial FSH dose will be chosen based on age, anti-Müllerian hormone (AMH) level, antral follicle count (AFC), and body mass index (BMI). The FSH dosage will be fixed during ovarian stimulation. Dydrogesterone (Duphaston, Abbott, USA) 20mg/day will start on the day of gonadotropin injection to the oocyte maturation trigger night.
  Interventions: Drug: Dydrogesterone 10 mg
- GnRH antagonist group (Active Comparator): GnRH antagonist group: Recombinant FSH 150-300 IU/day will be given from day 2 to day 4 of menstruation. The initial FSH dose will be chosen based on age, anti-Müllerian hormone (AMH) level, antral follicle count (AFC), and body mass index (BMI). The FSH dosage will be fixed during ovarian stimulation. Cetrorelix (Cetrotide, Merck, Germany) 0.25mg/day will be given from day 5 of stimulation by the oocyte maturation trigger day.
  Interventions: Drug: Cetrorelix 0.25 mg

INTERVENTIONS:
Drug: Dydrogesterone 10 mg — Dydrogesterone 10mg orally 2 times daily, starting on the day of gonadotropin injection to the oocyte maturation trigger night.
  Other Names: Duphaston
  Arms: Progestins Primed Ovarian stimulation group
Drug: Cetrorelix 0.25 mg — Cetrorelix 0.25mg is injected subcutaneously once a day. It is given from day 5 or day 6 of stimulation by the oocyte maturation trigger day.
  Other Names: Cetrotide
  Arms: GnRH antagonist group

SUMMARY:
This non-inferiority randomized controlled trial will be conducted at My Duc Hospital, Ho Chi Minh City, Vietnam.

This study compares the effectiveness of Progestin-Primed Ovarian stimulation versus GnRH protocol for ovarian stimulation in IVF treatment. Participants will be randomly assigned in a 1:1 ratio to receive Progestins or GnRH antagonists.

DETAILED DESCRIPTION:
Study Procedures

Participants will be randomized into two arms:

* PPOS group: Recombinant FSH 150-300 IU/day will start from day 2 to day 4 of menstruation. The initial FSH dose will be chosen based on age, anti-Müllerian hormone (AMH) level, antral follicle count (AFC), and body mass index (BMI). The FSH dosage will be fixed during ovarian stimulation. Dydrogesterone (Duphaston, Abbott, USA) 20mg/day will start on the day of gonadotropin injection to the oocyte maturation trigger night.
* GnRH antagonist group: Recombinant FSH 150-300 IU/day will be given from day 2 to day 4 of menstruation. The initial FSH dose will be chosen based on age, anti-Müllerian hormone (AMH) level, antral follicle count (AFC), and body mass index (BMI). The FSH dosage will be fixed during ovarian stimulation. Cetrorelix (Cetrotide, Merck, Germany) 0.25mg/day will be given from day 5 of stimulation by the oocyte maturation trigger day.

Follicular monitoring will start on the fifth or sixth day of ovarian stimulation and was performed every 3-5 days thereafter using transvaginal ultrasound to record the number of developing follicles. Measuring LH, estradiol, and progesterone serum levels will be performed on the fifth or sixth day of ovarian stimulation and oocyte maturation day (before the trigger injection). The FSH dosage will be fixed during ovarian stimulation. When more than two dominant follicles reach a diameter of at least 17mm, >= 50% diameter of remaining follicles cohort >=12 mm, the final stage of oocyte maturation will trigger using human chorionic gonadotropin (hCG; IVF-C 10.000 IU, LG Chem, Ltd., Korea or Ovitrelle Pen 250µg, Merck Serono S.p.A., Italy). In individuals who are at high risk for OHSS, GnRH agonist trigger 0.2mg (Diphereline 0.2mg, Ipsen Pharma, France) will given subcutaneously.

Transvaginal ultrasound-guided oocyte retrieval will be performed 34-36 hours after trigger, with the retrieval of all follicles exceeding 10mm in diameter. Oocyte fertilization will be carried out in vitro using ICSI. On the third day after fertilization, embryos will be evaluated for the degree of embryonic fragmentation, regularity, and number of blastomeres in accordance with the Istanbul consensus (Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology, 2011). Day 3 embryos will be cryopreserved or cultured until the blastocyst stage based on physician recommendation or patient references; viable blastocysts will then be cryopreserved on day 5 or day 6.

Endometrial preparation for frozen embryo transfer (FET) will be given using an exogenous steroid regimen from day 2 to day 4 of the menstrual cycle. Oral estradiol valerate (Progynova, Bayer Schering Pharma, Germany) 8mg/day will be given for 10-12 days. When endometrial thickness reaches ≥ 7mm, along with a triple-line pattern, micronized progesterone 800mg will be administered. FET will be performed three to five days after progesterone administration. There will be no more than 2 embryo(s) transfers each FET cycle. After FET, estradiol and progesterone supplementation will be continued for all participants until the day of taking the pregnancy test. Participants with a positive pregnancy test continued to receive oral estradiol valerate 8mg/day and micronized progesterone 800mg/day until the fetal heart appeared, and then only micronized progesterone 800mg will be used until 12 weeks of gestation.

All participants will be followed up per local protocol until outcomes are achieved.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18-40
* BMI ≤ 25kg/m2
* AMH > 1.2ng/mL or AFC >5
* Having indication for IVF treatment
* Agree to have frozen embryo(s) transfer
* Not participating in any other clinical trials
* Provision of written informed consent to participate

Exclusion Criteria:

* Undergoing IVF cycle with other protocols: Down-regulation, mild stimulation, Random start
* Oocyte donation cycles
* Undergoing vitrified oocyte accumulation
* Oocyte cryopreservation
* Cycle with PGT (Preimplatation genetic testing)
* Women with PCOS
* Women allergy to dydrogesterone, rFSH, GnRH antagonist

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 626 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy | At 10 weeks after embryo(s) placement
  defined as pregnancy with a detectable heart rate at 12 weeks gestation or beyond

SECONDARY OUTCOMES:
The incidence of premature LH surge | On the day having indication of oocyte maturation
  LH level of ≥ 10 mIU/mL occurring before the criteria of oocyte maturation administration is met
The incidence of premature progesterone elevation | On the day having indication of oocyte maturation
  A progesterone level of ≥1.0 ng/mL occurring before the criteria of oocyte maturation administration is met
Number of oocytes retrieved | On the oocyte(s) retrieval day
  The number of oocyte retrieved
Number of mature oocytes | On the oocyte(s) retrieval day
  The number of MII oocytes
Number of day 3 embryos | At 62-66 hours after ICSI
  The number of day 3 embryos
Number of day 5 embryos | At 112-116 hours after ICSI
  The number of day 5 embryos
Number of good quality day 3 embryos | At 62-66 hours after ICSI
  Number of grade 1 and grade 2 day 3 embryos (acccording to Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology, 2011)
Number of good quality day 5 embryos | At 112-116 hours after ICSI
  Number of grade 1 and grade 2 day 5 blastocysts (acccording to Alpha Scientists in Reproductive Medicine and ESHRE Special Interest Group of Embryology, 2011)
Number of frozen embryos | at 112-116 hours after ICSI
  the number of frozen embryos/blastocysts
Incidence of Ovarian hyperstimulation syndrome | At 2 weeks after trigger
  Ovarian hyperstimulation syndrome (OHSS) is a potentially lethal iatrogenic complication of the early luteal phase or/and early pregnancy after ovulation induction (OI) or ovarian stimulation (OS). OHSS was evaluated if symptoms were reported by the patient. OHSS was classified using the flow diagram developed by (Humaidan et al., 2016)
Positive ß-hCG test | At 2 weeks after embryo(s) placement
  Serum human chorionic gonadotropin level greater than 25 mIU/mL
Clinical pregnancy | at 6 weeks or more after the onset of last menstrual period
  diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of the last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ectopic pregnancy | at 6 weeks after the onset of last menstrual period
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology
Early miscarriage <12 weeks | At 12 weeks of gestation
  Spontaneous loss of intra-uterine pregnancy up to 12 weeks of gestation
Late miscariage 12-< 22 weeks | between 12 to 22 completed weeks of gestational age
  The spontaneous loss of an intra-uterine pregnancy between 12 to 22 completed weeks of gestational age
Live birth rate | At 22 weeks of gestation
  Defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heartbeat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is attached. A birth weight of 500 grams or more can be used if gestational age is unknown. Twins counted as one live birth.
Gestational age at birth | At birth
  Calculated by gestational age of all live births
Mode of delivery | At birth
  vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor)
Birth weight | At birth
  Weight of the newborn measured right after delivery
Very low birth weight | At birth
  Birth weight less than 1.500 g
Low birth weight | At birth
  Birth weight less than 2.500 g
High birth weight | At birth
  implies growth beyond an absolute birth weight, historically 4.000 g or 4.500 g, regardless of the gestational age
Very high birth weight | At birth
  Birth weight over than 4.500 g for women with diabetes, and a threshold of 5000 g for women without diabetes
Preterm birth | At birth
  defined as delivery at <24, <28, <32, <37 completed weeks. A birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Gestational diabetes mellitus | At 24 to 28 weeks of gestation
  a 75-g OGTT, with plasma glucose measurement when patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes.
  * Fasting: 92 mg/dL (5.1 mmol/L)
  * 1 h: 180 mg/dL (10.0 mmol/L)
  * 2 h: 153 mg/dL (8.5 mmol/L)
Hypertensive disorders of pregnancy | At 20 weeks of gestation or beyond
  Pregnancy-induced hypertension, pre-eclampsia, eclampsia and HELLP syndrome
Maternal mortality | From randomization to within 42 days of termination of pregnancy
  female deaths from any cause related to or aggravated by pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy
Major congenital abnormalities | From randomization to delivery
  Structural, functional, and genetic anomalies, that occur during pregnancy, and identified antenatally, at birth, or later in life, and require surgical repair of a defect, or are visually evident, or are life-threatening, or cause death. Any congenital anomaly will be included as followed definition of congenital abnormalities in Surveillance of Congenital Anomalies by Division of Birth Defects and Developmental Disabilities, NCBDDD, Centers for Disease Control and Prevention (2020)
NICU admission | at birth
  The admittance of the newborn to NICU
Reason for NICU admission | at birth
  Respiratory distress, Intraventricular Hemorrhage, Necrotizing enterocolitis, Sepsis
Neonatal mortality | within 28 days of birth
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between eight and 28 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Lan N Vuong, MD, PhD, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messinis IE. Ovarian feedback, mechanism of action and possible clinical implications. Hum Reprod Update. 2006 Sep-Oct;12(5):557-71. doi: 10.1093/humupd/dml020. Epub 2006 May 3. PMID 16672246
- [Background] Papanikolaou EG, Kolibianakis EM, Pozzobon C, Tank P, Tournaye H, Bourgain C, Van Steirteghem A, Devroey P. Progesterone rise on the day of human chorionic gonadotropin administration impairs pregnancy outcome in day 3 single-embryo transfer, while has no effect on day 5 single blastocyst transfer. Fertil Steril. 2009 Mar;91(3):949-52. doi: 10.1016/j.fertnstert.2006.12.064. Epub 2007 Jun 6. PMID 17555751
- [Background] Van Vaerenbergh I, Fatemi HM, Blockeel C, Van Lommel L, In't Veld P, Schuit F, Kolibianakis EM, Devroey P, Bourgain C. Progesterone rise on HCG day in GnRH antagonist/rFSH stimulated cycles affects endometrial gene expression. Reprod Biomed Online. 2011 Mar;22(3):263-71. doi: 10.1016/j.rbmo.2010.11.002. Epub 2010 Nov 13. PMID 21273126
- [Background] Droesch K, Muasher SJ, Brzyski RG, Jones GS, Simonetti S, Liu HC, Rosenwaks Z. Value of suppression with a gonadotropin-releasing hormone agonist prior to gonadotropin stimulation for in vitro fertilization. Fertil Steril. 1989 Feb;51(2):292-7. doi: 10.1016/s0015-0282(16)60493-4. PMID 2492234
- [Background] van Loenen AC, Huirne JA, Schats R, Hompes PG, Lambalk CB. GnRH agonists, antagonists, and assisted conception. Semin Reprod Med. 2002 Nov;20(4):349-64. doi: 10.1055/s-2002-36713. PMID 12536358
- [Background] Al-Inany HG, Youssef MA, Aboulghar M, Broekmans F, Sterrenburg M, Smit J, Abou-Setta AM. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2011 May 11;(5):CD001750. doi: 10.1002/14651858.CD001750.pub3. PMID 21563131
- [Background] Toftager M, Bogstad J, Bryndorf T, Lossl K, Roskaer J, Holland T, Praetorius L, Zedeler A, Nilas L, Pinborg A. Risk of severe ovarian hyperstimulation syndrome in GnRH antagonist versus GnRH agonist protocol: RCT including 1050 first IVF/ICSI cycles. Hum Reprod. 2016 Jun;31(6):1253-64. doi: 10.1093/humrep/dew051. Epub 2016 Apr 8. PMID 27060174
- [Background] Griesinger G, Schultz L, Bauer T, Broessner A, Frambach T, Kissler S. Ovarian hyperstimulation syndrome prevention by gonadotropin-releasing hormone agonist triggering of final oocyte maturation in a gonadotropin-releasing hormone antagonist protocol in combination with a "freeze-all" strategy: a prospective multicentric study. Fertil Steril. 2011 May;95(6):2029-33, 2033.e1. doi: 10.1016/j.fertnstert.2011.01.163. Epub 2011 Mar 2. PMID 21371705
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Wang Y, Chen Q, Wang N, Chen H, Lyu Q, Kuang Y. Controlled Ovarian Stimulation Using Medroxyprogesterone Acetate and hMG in Patients With Polycystic Ovary Syndrome Treated for IVF: A Double-Blind Randomized Crossover Clinical Trial. Medicine (Baltimore). 2016 Mar;95(9):e2939. doi: 10.1097/MD.0000000000002939. PMID 26945402
- [Background] Zhu X, Ye H, Fu Y. The Utrogestan and hMG protocol in patients with polycystic ovarian syndrome undergoing controlled ovarian hyperstimulation during IVF/ICSI treatments. Medicine (Baltimore). 2016 Jul;95(28):e4193. doi: 10.1097/MD.0000000000004193. PMID 27428219
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Vuong LN, Dang VQ, Ho TM, Huynh BG, Ha DT, Pham TD, Nguyen LK, Norman RJ, Mol BW. IVF Transfer of Fresh or Frozen Embryos in Women without Polycystic Ovaries. N Engl J Med. 2018 Jan 11;378(2):137-147. doi: 10.1056/NEJMoa1703768. PMID 29320655
- [Background] Shrestha D, La X, Feng HL. Comparison of different stimulation protocols used in in vitro fertilization: a review. Ann Transl Med. 2015 Jun;3(10):137. doi: 10.3978/j.issn.2305-5839.2015.04.09. PMID 26207230
- [Background] Ferin M, Rosenblatt H, Carmel PW, Antunes JL, Vande Wiele RL. Estrogen-induced gonadotropin surges in female rhesus monkeys after pituitary stalk section. Endocrinology. 1979 Jan;104(1):50-2. doi: 10.1210/endo-104-1-50. PMID 109276
- [Background] Leroy I, d'Acremont M, Brailly-Tabard S, Frydman R, de Mouzon J, Bouchard P. A single injection of a gonadotropin-releasing hormone (GnRH) antagonist (Cetrorelix) postpones the luteinizing hormone (LH) surge: further evidence for the role of GnRH during the LH surge. Fertil Steril. 1994 Sep;62(3):461-7. doi: 10.1016/s0015-0282(16)56932-5. PMID 8062939